CLINICAL TRIAL: NCT00590707
Title: A Strategy to Reduce the Incidence of Post-Operative Delirium in Elderly Patients
Brief Title: Post-Operative Delirium in Elderly Surgical Patients
Acronym: STRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NA_00041873; ACCM Delirium 3; R01AG033615 (NIH)
Record Dates: First submitted 2007-12-28; First posted 2008-01-11 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Hip Fractures; Delirium
Keywords: Hip fractures; Femoral neck fractures; Trochanteric fractures; Intertrochanteric fractures; Subtrochanteric fractures; Delirium; Confusion
MeSH Terms: conditions — Hip Fractures; Delirium; Femoral Neck Fractures; Confusion | interventions — Conscious Sedation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Deeper sedation (Active Comparator): Patients randomly assigned to this arm will receive enough sedative drugs to keep their level of awareness during the hip fracture repair, as measured by the use of the Observer's Assessment of Awareness/Sedation Scale (OAA/S), at an OAA/S score of 0. This is the "deeper sedation" arm.
  Interventions: Device: Deeper sedation
- Moderate sedation (Active Comparator): Patients randomly assigned to this arm will receive enough sedative drugs to keep their level of awareness during the hip fracture repair, as measured by the use of the Observer's Assessment of Awareness/Sedation Scale (OAA/S), at an OAA/S score of 4-5. This is the "moderate sedation" arm.
  Interventions: Device: Moderate sedation

INTERVENTIONS:
Device: Deeper sedation — The depth of sedation, as measured by the use of the Observer's Assessment of Awareness/Sedation Scale (OAA/S), will be maintained at an OAA/S score of 0.
  Other Names: Observer's Assessment of Awareness/Sedation Scale (OAA/S)
  Arms: Deeper sedation
Device: Moderate sedation — The depth of sedation, as measured by the use of the Observer's Assessment of Awareness/Sedation Scale (OAA/S), will be maintained at an OAA/S score of 4-5.
  Other Names: Observer's Assessment of Awareness/Sedation Scale (OAA/S)
  Arms: Moderate sedation

SUMMARY:
This research is being done to see what effects sedative drugs during surgery have on peoples' thinking processes after they wake up.

DETAILED DESCRIPTION:
We give sedative drugs to patients having spinal anesthesia so they are "asleep" (sedated) while we are fixing their broken hips. The spinal anesthesia provides pain relief at the site of surgery, while the sedative drugs keep people "asleep" during the procedure. We want to find out whether the amount of sedation we give might (1) make patients be confused when they wake up or (2) have anything to do with how well patients can do their ordinary daily routines a few months after their surgery.

ELIGIBILITY:
Inclusion Criteria:

* is 65 years of age or older at admission;
* has surgical treatment of a traumatic hip fracture;
* has participating surgeon;
* has Mini-Mental Status Exam score of 15 or higher;
* able to read/write/speak/hear/understand English;
* gives informed consent;
* receives spinal anesthesia

Exclusion Criteria:

* receives general anesthesia;
* does not write/write/speak/hear/understand English;
* has severe chronic obstructive pulmonary disease (COPD);
* has severe congestive heart failure (CHF);
* has Mini-Mental Status Exam score less than 15;
* declines to give informed consent;
* age less than 65 years at admission;
* attending surgeon does not participate in study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick E. Sieber, MD, Principal Investigator — Dept. of Anesthesiology and Critical Care Medicine, School of Medicine, The Johns Hopkins University
Locations (1):
- The Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Sieber F, Neufeld KJ, Gottschalk A, Bigelow GE, Oh ES, Rosenberg PB, Mears SC, Stewart KJ, Ouanes JP, Jaberi M, Hasenboehler EA, Wang NY. Depth of sedation as an interventional target to reduce postoperative delirium: mortality and functional outcomes of the Strategy to Reduce the Incidence of Postoperative Delirium in Elderly Patients randomised clinical trial. Br J Anaesth. 2019 Apr;122(4):480-489. doi: 10.1016/j.bja.2018.12.021. Epub 2019 Feb 4. PMID 30857604
- [Derived] Sieber FE, Neufeld KJ, Gottschalk A, Bigelow GE, Oh ES, Rosenberg PB, Mears SC, Stewart KJ, Ouanes JP, Jaberi M, Hasenboehler EA, Li T, Wang NY. Effect of Depth of Sedation in Older Patients Undergoing Hip Fracture Repair on Postoperative Delirium: The STRIDE Randomized Clinical Trial. JAMA Surg. 2018 Nov 1;153(11):987-995. doi: 10.1001/jamasurg.2018.2602. PMID 30090923
- [Derived] Sieber FE, Zakriya KJ, Gottschalk A, Blute MR, Lee HB, Rosenberg PB, Mears SC. Sedation depth during spinal anesthesia and the development of postoperative delirium in elderly patients undergoing hip fracture repair. Mayo Clin Proc. 2010 Jan;85(1):18-26. doi: 10.4065/mcp.2009.0469. PMID 20042557

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Deeper Sedation | Moderate Sedation
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deeper Sedation | Moderate Sedation | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 82 (7) | 82 (8) | 82 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 72 | 146
  Male | 26 | 28 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 97 | 97 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Presence of Delirium as Assessed by the Confusion Assessment Method
Description: The presence of delirium is assessed by the confusion assessment method (CAM), during postoperative Day 1 to Day 5 or up to hospital discharge, whichever occurs first. The CAM consists of 4 features: 1-Onset, 2-Inattention, 3-Disorganized thinking, and 4-altered level of consciousness. The diagnosis of delirium by CAM is based on the presence of features 1 and 2, and either 3 or 4.
Time Frame: Postoperative days up to hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Deeper Sedation | Moderate Sedation
Number analyzed (Participants) | 100 | 100
Participants | 39 | 34

2. Secondary Outcome: Change in Functional Status
Description: Ability to perform Activities of Daily Living (ADL) using 6-point Katz activities of daily living scale, assessed at 12 months post-op. The range of the Katz activities of daily living scale is from 0-6, 0 is worse and 6 is best.
Time Frame: 12 months post-operative
Population: ADL score at 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deeper Sedation | Moderate Sedation
Number analyzed (Participants) | 100 | 100
units on a scale | 4.2 (1.5) | 4.1 (1.6)

3. Secondary Outcome: Mortality
Description: death occurring during follow-up period, in one year post-op.
Time Frame: 12 months post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Deeper Sedation | Moderate Sedation
Number analyzed (Participants) | 100 | 100
Participants | 14 | 14

4. Secondary Outcome: Number of Participants With the Presence of Delirium at 1 Month as Assessed by the Confusion Assessment Method
Description: The presence of delirium is assessed by the confusion assessment method (CAM), after 1 month postoperative. The CAM consists of 4 features: 1-Onset, 2-Inattention, 3-Disorganized thinking, and 4-altered level of consciousness. The diagnosis of delirium by CAM is based on the presence of features 1 and 2, and either 3 or 4.
Time Frame: 1 month (30 days) post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Deeper Sedation | Moderate Sedation
Number analyzed (Participants) | 100 | 100
Participants | 3 | 1

5. Secondary Outcome: Clinical Dementia Rating Sum of Boxes (CDR-SOB) Score
Description: Clinical Dementia Rating consists of 6 domains ("boxes") of function: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain ("box") is rated on a 5-point scale (0= no impairment, 0.5=questionable impairment, 1= mild impairment, 2= moderated impairment, 3= severe impairment. The CDR-SOB score is a sum of these ratings, for a total Sum of boxes ranging from 0-18, where 0=cognitively intact. Increasing sum of boxes score is associated with greater cognitive impairment.
Time Frame: 12 months post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deeper Sedation | Moderate Sedation
Number analyzed (Participants) | 100 | 100
units on a scale | 2.0 (3.0) | 2.0 (3.0)

ADVERSE EVENTS:
Time Frame: 1 year
Description: definitions are same as clinical trials.gov definitions
Arm/Group | Deeper Sedation | Moderate Sedation
All-Cause Mortality (participants affected / at risk) | 14/100 | 14/100
Serious Adverse Events (participants affected / at risk) | 15/100 | 14/100
Other Adverse Events (participants affected / at risk) | 69/100 | 69/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deeper Sedation (N=100) | Moderate Sedation (N=100)
cardiaovascular postop complications (Cardiac disorders) | 3 (3) | 3 (3)
wound (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
cns (Nervous system disorders) | 2 (2) | 3 (3)
urinary tract (Renal and urinary disorders) | 1 (1) | 1 (1)
orthopedic (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
other postop (Surgical and medical procedures) | 5 (5) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deeper Sedation (N=100) | Moderate Sedation (N=100)
urinary tract (Renal and urinary disorders) | 37 (37) | 42 (42)
wound (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
respiratory (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
cns (Nervous system disorders) | 0 (0) | 1 (1)
cardiovascualr (Cardiac disorders) | 9 (9) | 10 (10)
orthopedic (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
other postop (Surgical and medical procedures) | 16 (16) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT00590707/Prot_SAP_000.pdf